CLINICAL TRIAL: NCT06037473
Title: A Real-world Study of the Efficacy and Safety of PEGylated Recombinant Human Growth Hormone Injection in the Treatment of Short Stature in Chinese Children From the Global Registry for Novel Therapies For Rare Bone or Endocrine Conditions
Brief Title: The Efficacy and Safety of PEGylated GH for the Treatment of Short Stature in Chinese Children-GLOBE Reg
Status: Recruiting | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Chunxiu Gong, Principal Investigator, Beijing Children's Hospital
Other Study IDs: Gensci-LAGH-23003
Record Dates: First submitted 2023-08-15; First posted 2023-09-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Growth Hormone Treatment; Growth Disorders
MeSH Terms: conditions — Growth Disorders | interventions — polyethylene glycol-recombinant human growth hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- growth hormone deficiency(GHD): Growth hormone deficiency (GHD) is a rare and treatable condition that causes short height in children and metabolic issues in adults.
  Interventions: Drug: Polyethylene glycol recombinant human growth hormone injection
- Idiopathic short stature (ISS): Idiopathic short stature is a condition in which the height of the individual is more than 2 SD below the corresponding mean height for a given age, sex and population, in whom no identifiable disorder is present.
  Interventions: Drug: Polyethylene glycol recombinant human growth hormone injection
- small for gestational age (SGA): Small for gestational age (SGA) is defined as a birth weight of less than 10th percentile for gestational age.
  Interventions: Drug: Polyethylene glycol recombinant human growth hormone injection
- Turner Syndrome (TS): Turner syndrome, a condition that affects only females, results when one of the X chromosomes (sex chromosomes) is missing or partially missing.
  Interventions: Drug: Polyethylene glycol recombinant human growth hormone injection
- others: others who with the height of the individual is more than 2 SD below the corresponding mean height for a given age, sex and population.
  Interventions: Drug: Polyethylene glycol recombinant human growth hormone injection

INTERVENTIONS:
Drug: Polyethylene glycol recombinant human growth hormone injection — 0.1-0.3mg/kg.w

SUMMARY:
In order to further observe the long-term safety and effectiveness of real-world polyethylene glycol-recombinant human growth hormone(PEG-rhGH) treatment of GHD, idiopathic short stature, and SGA in children, explore and analyze the factors affecting the efficacy of PEG-rhGH and the height prediction model after treatment, etc., collect and analyze more scientifically and rationally, and understand the situation of real-world PEG-GH treatment. A database registration study was developed.

DETAILED DESCRIPTION:
A database registration study was developed to retrospectively analyze the efficacy and safety of polyethylene glycol recombinant human growth hormone injection in the treatment of slow growth in children caused by endogenous growth hormone deficiency, idiopathic short stature, Turner syndrome, etc., and to further prospectively follow up and monitor. In order to participate in the global real-world use of long-acting growth hormone, all data from this study were uploaded to the Global Registry of New Therapies for Rare Endocrine Diseases and Bone Disorders (GloBE-Reg) platform.

ELIGIBILITY:
Inclusion Criteria:

Patients with endogenous growth hormone deficiency, Turner Syndrome, SGA, idiopathic short stature, etc. treated with polyethylene glycol recombinant human growth hormone injection

Exclusion Criteria:

Patients with serious heart and lung, blood system, malignant tumors and other diseases or systemic infections, immune function is low and Persons with mental illness;

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The height of the patients was below 2 stadard deviation below average. The patients were diagosesed as endogenous growth hormone deficiency, TS, SGA, ISS, etc. and treated with polyethylene glycol recombinant human growth hormone injection
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
the change in height standard deviation score | 3-10years
  final adult height standard deviation score- height standard deviation score before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bingyan Cao, Dr., Principal Investigator — Beijing Children's Hospital
Locations (1):
- Department of Endocrinology, Genetics, Metabolism, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided